CLINICAL TRIAL: NCT02038933
Title: A Single-Arm, Open-Label, Phase 2 Study of Nivolumab (BMS-936558) in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) After Failure of Autologous Stem Cell Transplant (ASCT) or After Failure of At Least Two Prior Multi-Agent Chemotherapy Regimens in Subjects Who Are Not Candidates for ASCT
Brief Title: Study of Nivolumab in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) That Have Either Failed or Are Not Eligible for Autologous Stem Cell Transplant (CheckMate 139)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-139; 2013-003621-28 (EudraCT Number)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma. Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nivolumab (3 mg/kg) (Experimental): Nivolumab 3 mg/kg solution intravenously every 2 weeks until progression or unacceptable toxicity
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
  Other Names: BMS-936558

SUMMARY:
The purpose of this study is to determine whether Nivolumab is effective in the treatment of DLBCL in patients that have failed or are ineligible for ASCT

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Confirmation of relapsed or refractory DLBCL or transformed lymphoma (TL)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 -1
* At least one lesion that measures >1.5 cm
* Prior therapy and screening lab criteria must be met
* Appropriate contraceptive measures must be taken

Exclusion Criteria:

* Known central nervous system (CNS) lymphoma
* History of interstitial lung disease, prior malignancy, active autoimmune disease, positive test for hepatitis B or hepatitis C virus
* Prior allogeneic stem cell transplant (SCT), chest radiation ≤ 24 weeks from study drug, ≥1000 mg of Carmustine Bis-chloroethylnitrosourea (BCNU) as part of pre-transplant conditioning regimen, prior treatment with drug targeting T-cell costimulation or immune checkpoint pathways
* Women who are breastfeeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (44):
- United States (10):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Division Of Hematology & Oncology Ctr. For Health Sciences, Los Angeles, California
  - Winship Cancer Center, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center (Cumc), New York, New York
  - Weill Cornell Medical College, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (3):
  - Local Institution, Waratah, New South Wales
  - Local Institution, Woodville, South Australia
  - Local Institution, Heidelberg, Victoria
- Belgium (3):
  - Local Institution, B-leuven
  - Local Institution, Brussels
  - Local Institution, Ghent
- Canada (2):
  - Local Institution, Montreal, Quebec
  - Local Institution, Montreal
- France (4):
  - Local Institution, Créteil
  - Hopital Saint Eloi, Montpellier
  - Local Institution, Pierre-Bénite
  - Local Institution, Rennes
- Germany (4):
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Homburg
  - Local Institution, Ulm
- Italy (5):
  - Local Institution, Bergamo
  - Local Institution, Bologna
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Roma
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Rotterdam
  - Local Institution, Utrecht
- Local Institution, Singapore, Singapore
- Spain (4):
  - Local Institution, Hospitalet Llobregat- Barcelona
  - Local Institution, Madrid
  - Hospital Universitario La Paz, Madrid
  - Local Institution, Salamanca
- Sweden (2):
  - Local Institution, Gothenburg
  - Local Institution, Lund
- United Kingdom (3):
  - Local Institution, Southampton, Hampshire
  - Local Institution, Withington, Manchester
  - Local Institution, Sutton, Surrey

REFERENCES:
- [Derived] Ansell SM, Minnema MC, Johnson P, Timmerman JM, Armand P, Shipp MA, Rodig SJ, Ligon AH, Roemer MGM, Reddy N, Cohen JB, Assouline S, Poon M, Sharma M, Kato K, Samakoglu S, Sumbul A, Grigg A. Nivolumab for Relapsed/Refractory Diffuse Large B-Cell Lymphoma in Patients Ineligible for or Having Failed Autologous Transplantation: A Single-Arm, Phase II Study. J Clin Oncol. 2019 Feb 20;37(6):481-489. doi: 10.1200/JCO.18.00766. Epub 2019 Jan 8. PMID 30620669
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 121 participants entered the treatment period.
Groups:
- Nivolumab 3mg/kg: Nivolumab 3mg/kg IV Q2W for participants who failed autologous stem cell transplant (ASCT) or who were ineligible for ASCT
Period: Overall Study
Arm/Group | Nivolumab 3mg/kg
Started | 121
Completed | 0
Not Completed | 121
Not completed — Disease progression | 104
Not completed — Study drug toxicity | 6
Not completed — Adverse event unrelated to study drug | 6
Not completed — Participant request to discontinue treatment | 2
Not completed — Lost to Follow-up | 1
Not completed — Other reasons | 2

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- ASCT-failed: Participants who failed Autologous stem cell transplant (ASCT), treated with Nivolumab 3 mg/Kg Q2W
- ASCT-ineligible: Participants who were ineligible for Autologous stem cell transplant (ASCT), treated with Nivolumab 3 mg/Kg Q2W
- Total: Total of all reporting groups
Arm/Group | ASCT-failed | ASCT-ineligible | Total
Number analyzed (Participants) | 87 | 34 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.94) | 66.4 (12.98) | 61.1 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 13 | 44
  Male | 56 | 21 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 44 | 20 | 64
  Unknown or Not Reported | 41 | 13 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 71 | 31 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Independent Radiologic Review Committee (IRRC) Assessment
Description: ORR is defined as the percentage of participants with a Best Overall Response (BOR) of Complete Remission (CR) or Partial Remission (PR), according to the 2007 revised International Working Group (IWG) Criteria for Malignant Lymphoma, , based on IRRC assessment. CR= Disappearance of all evidence of disease, confirmed by PET scan; PR= Regression of measurable disease and no emergence of new sites
Time Frame: From first dose until date of documented disease progression or subsequent therapy, whichever occurs first (assesed up to April 2016, approximately 25 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | ASCT-failed | ASCT-ineligible
Number analyzed (Participants) | 87 | 34
Percent of participants | 10.3 [4.8 to 18.7] | 2.9 [0.1 to 15.3]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first response (Complete Response (CR) or Partial Response (PR)) to the date of initial objectively documented progression as determined using the 2007 revised IWG Criteria for Malignant Lymphoma, based on Independent Radiology Review Committee (IRRC) assessment, or death due to any cause, whichever occurs first. CR= Disappearance of all evidence of disease, confirmed by PET scan; PR= Regression of measurable disease and no emergence of new sites.
Time Frame: From date of first response to the date of documented disease progression or death, whichever occurs first (up to approximately 18 months)
Population: All participants with CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ASCT-failed | ASCT-ineligible
Number analyzed (Participants) | 9 | 1
Months | 11.43 [2.53 to 17.15] | 8.34 [NA to NA] — 95% CI was not calculated as there was only one participant analyzed in this arm.

3. Secondary Outcome: Complete Remission Rate
Description: Complete Remission Rate is defined as the percentage of participants with a Best Overall Response (BOR) of Complete Response (CR) according to the 2007 revised IWG Criteria for Malignant Lymphoma, based on Independent Radiology Review Committee (IRRC) assessment. CR= Disappearance of all evidence of disease, confirmed by PET scan.
Time Frame: From date of first dose to study completion (up to approximately 78 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | ASCT-failed | ASCT-ineligible
Number analyzed (Participants) | 87 | 34
Percent of participants | 3.4 [0.7 to 9.7] | 0 [0 to 10.3]

4. Secondary Outcome: Duration of Complete Remission
Description: The duration of Complete Remission is defined as the time from first documentation of Complete Response (CR) (which is the date of first negative FDG-PET scan or the date of first documentation of no disease involvement in the bone marrow [if required], whichever occurs later) to the date of initial objectively documented progression as determined using the 2007 IWG criteria, based on Independent Radiology Review Committee (IRRC) assessment, or death due to any cause, whichever occurs first.
  CR= Disappearance of all evidence of disease, confirmed by PET scan.
Time Frame: From time of first documentation of CR to the date of initial documented disease progression or death due to any cause, whichever occurs first (up approximately 14 months)
Population: All participants with CR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ASCT-failed | ASCT-ineligible
Number analyzed (Participants) | 3 | 0
Months | NA [11.17 to NA] — Median and Upper Limit were not reached due to insufficient number of participants with CR |

5. Secondary Outcome: Partial Remission Rate
Description: Partial Remission rate is defined as the percentage of participants with a Best Overall Response (BOR) of Partial Response (PR) according to the 2007 revised IWG Criteria for Malignant Lymphoma, based on Independent Radiology Review Committee (IRRC) assessment. PR= Regression of measurable disease and no emergence of new sites.
Time Frame: From date of first dose to study completion (up to approximately 78 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | ASCT-failed | ASCT-ineligible
Number analyzed (Participants) | 87 | 34
Percent of participants | 6.9 [2.6 to 14.4] | 2.9 [0.1 to 15.3]

6. Secondary Outcome: Duration of Partial Remission
Description: Duration of Partial Remission is defined as the time from first documentation of Partial Response (PR) to the date of initial objectively documented progression as determined using the 2007 IWG criteria, based on Independent Radiology Review Committee (IRRC) assessment, or death due to any cause, whichever occurs first.
  PR= Regression of measurable disease and no emergence of new sites.
Time Frame: From date of first documentation of PR to date of disease progression or death due to any cause, whichever occurs first (up to approximately 12 months)
Population: All participants with PR
Measure: Median (Full Range); unit: Months
Arm/Group | ASCT-failed | ASCT-ineligible
Number analyzed (Participants) | 6 | 1
Months | 6.64 [2.4 to 11.4] | 8.34 [8.34 to 8.34]

7. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) is defined as the time from first dosing date to the date of the first documented progression, as determined by an Independent Radiology Review Committee (IRRC) according to the 2007 revised IWG Criteria for Malignant Lymphoma, or death due to any cause, whichever occurs first.
Time Frame: From date of first dose to date of documented disease progression or death due to any cause, whichever occurs first (up to approximately 2 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ASCT-failed | ASCT-ineligible
Number analyzed (Participants) | 87 | 34
Months | 1.87 [1.71 to 1.87] | 1.41 [1.15 to 1.81]

8. Secondary Outcome: Objective Response Rate (ORR) Per Investigator Assessment
Description: ORR is defined as the percentage of participants with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR), according to investigator assessment.
  CR= Disappearance of all evidence of disease, confirmed by PET scan; PR= Regression of measurable disease and no emergence of new sites.
Time Frame: From first dose until date of documented disease progression or subsequent therapy, whichever occurs first (up to approximately 30 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | ASCT-failed | ASCT-ineligible
Number analyzed (Participants) | 87 | 34
Percent of participants | 19.5 [11.8 to 29.4] | 2.9 [0.1 to 15.3]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of first dose to study completion (up to approximately 79 months). Serious Adverse events and other adverse events were assessed from date of first dose to 100 days following date of last dose (up to approximately 66 months)
Arm/Group | NIVOLUMAB 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 98/121
Serious Adverse Events (participants affected / at risk) | 83/121
Other Adverse Events (participants affected / at risk) | 109/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB 3 mg/kg (N=121)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Eye swelling (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Oesophageal perforation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Facial pain (General disorders) | 1
General physical health deterioration (General disorders) | 3
Localised oedema (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 4
Swelling face (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 2
Neutropenic sepsis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pneumonia bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Transaminases increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 1
Morphoea (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
IIIrd nerve paralysis (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Renal impairment (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB 3 mg/kg (N=121)
Anaemia (Blood and lymphatic system disorders) | 32
Neutropenia (Blood and lymphatic system disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Abdominal pain (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 27
Diarrhoea (Gastrointestinal disorders) | 25
Dry mouth (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 41
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 23
Asthenia (General disorders) | 8
Fatigue (General disorders) | 49
Oedema peripheral (General disorders) | 17
Pyrexia (General disorders) | 29
Nasopharyngitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 9
Aspartate aminotransferase increased (Investigations) | 8
Blood creatinine increased (Investigations) | 13
Decreased appetite (Metabolism and nutrition disorders) | 23
Hypercalcaemia (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Headache (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Night sweats (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT02038933/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT02038933/SAP_001.pdf